CLINICAL TRIAL: NCT02509897
Title: Cardiorespiratory, Metabolic and Immunoregulatory Response to Hypoxia in Multiple Sclerosis Patients: A Pilot Study
Brief Title: Normobaric Hypoxic Training and Multiple Sclerosis
Acronym: MS_EPOXI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Anja Maehler, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EpoxiMet
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: Hypoxia training; Activity energy expenditure; Immunoregulation; Energy Metabolism; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxic training (Active Comparator): Endurance training
  Interventions: Other: Hypoxic training
- Normoxic training (Placebo Comparator): Endurance training
  Interventions: Other: Normoxic training

INTERVENTIONS:
Other: Hypoxic training — Hypoxic training 3 times per week four four weeks
  Arms: Hypoxic training
Other: Normoxic training — Normoxic training 3 times per week four four weeks
  Arms: Normoxic training

SUMMARY:
To study the effects of normobaric hypoxic training on cardiorespiratory fitness, resting, postprandial and exercise activity energy expenditure, immunoregulatory functions and serum erythropoietin levels in relapsing-remitting multiple sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* stable immunomodulatory therapy
* expanded disability status scale score < 4.5
* body mass index 18.5 - 29.9 kg/m2

Exclusion Criteria:

* clinically relevant heart, lung, liver, and kidney diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Activity energy expenditure measured by indirect calorimetry (respiratory chamber) | Change from baseline at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental & Clinical Research Center, Berlin, Germany

REFERENCES:
- [Result] Mahler A, Balogh A, Csizmadia I, Klug L, Kleinewietfeld M, Steiniger J, Susnjar U, Muller DN, Boschmann M, Paul F. Metabolic, Mental and Immunological Effects of Normoxic and Hypoxic Training in Multiple Sclerosis Patients: A Pilot Study. Front Immunol. 2018 Nov 29;9:2819. doi: 10.3389/fimmu.2018.02819. eCollection 2018. PMID 30555484
- See also: Results publication — http://www.frontiersin.org/articles/10.3389/fimmu.2018.02819/full